CLINICAL TRIAL: NCT04833842
Title: The Effect of Pre-Birth Program Developed Based on Health Belief Model on Fear of Birth, Birth Self-Efficacy, Birth Process and Perception in Primigravida Pregnant Women
Brief Title: Childbirth Preparation Program Developed Based on Health Belief Model
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Cumhuriyet University (Other)
Responsible Party: Principal Investigator, Bi̇rnur Yeşi̇ldağ Çeli̇k, lecturer, Cumhuriyet University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: SİVAS CUMHURİYET ÜNİVERSİTESİ
Record Dates: First submitted 2021-03-31; First posted 2021-04-06 (Actual); Last update posted 2021-04-06 (Actual); Status verified 2021-04

CONDITIONS: Fear of Childbirth; Self-efficacy
Keywords: motivational interviewing; childbirth training; fear of childbirth,; self-efficacy; primigravida women

STUDY DESIGN:
Intervention Model Description: This study is a randomized controlled trial.
Who Masked: Participant, Outcomes Assessor
Masking Description: In the study, the single blinding method, in which the participants are blinded, will be used. A placebo-controlled approach will be used in the control group (website training group) so that the participants in the groups do not know which group they are in. In the research, the statistician who also evaluates the outputs and performs data analysis will be blinded.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Web-based birth preparation program supported by motivational interview (Experimental): A web-based childbirth preparation program prepared based on the Health Belief Model and supported by motivational interviews will be applied to primigravida women in the initiative group.
  Interventions: Other: Web-based childbirth preparation program developed based on health belief model and supported by motivational interview
- web-based birth preparation program (Experimental): A web-based birth preparation program based on the Health Belief Model will be applied to primigravida women in the control group.
  Interventions: Other: Web-based childbirth preparation program based on health belief model

INTERVENTIONS:
Other: Web-based childbirth preparation program developed based on health belief model and supported by motivational interview — In the three-month study, primigravida women in the initiative group will be given a web-based childbirth preparation program, which is prepared based on the Health Belief Model and supported by motivational interviews. Before starting the training program, pre-test will be applied to pregnant women and a five-week program will be implemented. A final test will be applied at the end of the program. The birth process will be evaluated immediately after the pregnant women give birth.
  Arms: Web-based birth preparation program supported by motivational interview
Other: Web-based childbirth preparation program based on health belief model — In the three-month study, a web-based childbirth preparation program based on the Health Belief Model will be applied to primigravida women in the control group. Before starting the training program, pre-test will be applied to pregnant women and a five-week program will be implemented. A final test will be applied at the end of the program. The birth process will be evaluated immediately after the pregnant women give birth.
  Arms: web-based birth preparation program

SUMMARY:
Pregnants who underwent a web-based preparation for labor program, which was developed based on the health belief model and supported by motivational interviews, had a higher perception of birth self-efficacy than those who did not pass.

Pregnant women who underwent a web-based preparation for labor program, which was developed based on a health belief model and supported by motivational interviews, had a more positive perception of birth than those who did not pass.

The level of fear experienced at birth is lower in pregnant women who underwent a web-based preparation for labor program, which was developed based on the health belief model and supported by motivational interviews.

The frequency of voluntary cesarean delivery is lower in pregnant women who undergo a web-based preparation for labor program, which is developed based on the health belief model and supported by motivational interviews.

The frequency of episiotomy is lower in pregnant women who undergo a web-based preparation for labor program, which is developed based on a health belief model and supported by motivational interviews.

Induction frequency is lower in pregnant women who underwent a web-based preparation for labor program, which was developed based on the health belief model and supported by motivational interviews, than those who did not pass.

Pregnants who underwent a web-based preparation program for labor, which was developed based on the health belief model and supported by motivational interviews, had a shorter delivery period than those who did not pass.

DETAILED DESCRIPTION:
In the three-month study, a web-based childbirth preparation program will be applied to primigravida women in the initiative group, based on the Health Belief Model and supported by motivational interviews. Training will take five weeks. Beginning from the 30th week of pregnancy, pregnant women will be asked to read the first part of the website and a suitable time will be determined for a motivational interview by calling the phone within that week. All applications of pregnant women related to the website will be evaluated. At the specified time, pregnant women will be taken to motivational interview training based on the Health Belief Model and the trainings will be carried out individually and online. A web-based birth preparation program based on the Health Belief Model will be applied to primigravida women in the control group. Training will take five weeks. Beginning from the 30th week of pregnancy, pregnant women will be asked to read the first part of the website. All applications of pregnant women related to the website will be evaluated.

ELIGIBILITY:
Inclusion Criteria:

* Between the ages of 18-35,
* At least a primary school graduate,
* According to the last menstrual period or the results of ultrasonography of pregnant women who do not know the last menstrual period, who are in the 28-30 weeks of pregnancy,
* Primigravida,
* Live single pregnancy,
* Without any obstacle to give birth through normal vaginal way,
* No specified cesarean indication or risk factors that would adversely affect normal delivery (Heart disease, placenta previa, oligohydramnios, preeclampsia, anhydramnios, diabetes, epilepsy),
* Not pregnant as a result of infertility treatment,
* The state anxiety scale average score is below 60,
* Edinburgh Postpartum Depression Scale average score of 12 or below,
* Residing within the provincial borders of Sivas,
* Internet at home,
* Able to use a computer or mobile phone,
* They are pregnant women who agree to participate in the research.

Exclusion Criteria:

* Participants in the birth preparation class

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — primigravida pregnant women
Enrollment: 74 (Estimated)
Dates: Start 2021-04-15 (Estimated); Primary Completion 2021-06-15 (Estimated); Study Completion 2021-07-30 (Estimated)

PRIMARY OUTCOMES:
has an effect on the fear of childbirth fear of birth birth self-efficacy | 3 months
  Wijma Birth Expectation / Experience Scale Version A: It is a scale consisting of 33 items. The answers in the scale are numbered from 0 to 5, and are in six-point Likert type. Zero is expressed as "completely" and 5 as "nothing". While the minimum score on the scale is 0, the maximum score is 165. A high item total score indicates a high level of fear. Eighty-five and above points indicate clinical level fear.
has an impact on birth self-efficacy | 3 months
  Short Version of the Self-Efficacy Scale in Labor: Each sub-dimension of the scale consists of two sub-dimensions, and consists of 16 questions. The lowest score to be obtained from the scale sub-dimensions is 16 and the highest score is 160. The lowest total score that can be obtained from the scale is 32, and the total highest score is 320. High scores to be obtained from the scale indicate that pregnant women have high levels of self-efficacy in labor.
has an effect on birth health belief | 3 months
  Birth Health Belief Scale: The scale consists of 34 items and has five sub-dimensions. According to the subscales of the scale, the average "self-efficacy and motivation perception" is high 3.810 ± 1.409 (Min = 1; Max = 5), the average "benefit and motivation perception" is very high 4.368 ± 0.909 (Min = 1.75; Max = 5), "sensitivity perception of perception high 3,500 ± 1,502 (Min = 1; Max = 5), "caring / seriousness perception" average high 3,441 ± 1,600 (Min = 1; Max = 5), average "obstacle perception" 3,071 ± 1,508 (Min = 1; Max = 5).

CONTACTS AND LOCATIONS:
Overall Officials: BİRNUR YEŞİLDAĞ ÇELİK, Lecturer, Principal Investigator — SİVAS CUMHURİYET UNIVERSITY; ZEHRA GÖLBAŞI, Prof. Dr, Study Director — LOKMAN HEKİM UNIVERSITY
Locations (1):
- Sivas Cumhuriyet Üniversitesi, Sivas, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
All IPD collected will share
Supporting Information: Study Protocol
Time Frame: starts 1 month after broadcast
Access Criteria: all people have access.

REFERENCES:
- [Background] Artieta-Pinedo I, Paz-Pascual C, Grandes G, Remiro-Fernandezdegamboa G, Odriozola-Hermosilla I, Bacigalupe A, Payo J. The benefits of antenatal education for the childbirth process in Spain. Nurs Res. 2010 May-Jun;59(3):194-202. doi: 10.1097/NNR.0b013e3181dbbb4e. PMID 20421842
- [Background] Munkhondya BMJ, Munkhondya TE, Chirwa E, Wang H. Efficacy of companion-integrated childbirth preparation for childbirth fear, self-efficacy, and maternal support in primigravid women in Malawi. BMC Pregnancy Childbirth. 2020 Jan 21;20(1):48. doi: 10.1186/s12884-019-2717-5. PMID 31964346
- [Background] Byrne J, Hauck Y, Fisher C, Bayes S, Schutze R. Effectiveness of a Mindfulness-Based Childbirth Education pilot study on maternal self-efficacy and fear of childbirth. J Midwifery Womens Health. 2014 Mar-Apr;59(2):192-7. doi: 10.1111/jmwh.12075. Epub 2013 Dec 10. PMID 24325752
- [Background] Toohill J, Fenwick J, Gamble J, Creedy DK, Buist A, Turkstra E, Ryding EL. A randomized controlled trial of a psycho-education intervention by midwives in reducing childbirth fear in pregnant women. Birth. 2014 Dec;41(4):384-94. doi: 10.1111/birt.12136. Epub 2014 Oct 9. PMID 25303111